CLINICAL TRIAL: NCT07357025
Title: Longitudinal Resting-State fMRI Assessment of Brain Functional Connectivity in Patients With Trigeminal Neuralgia Treated by Gamma Knife Radiosurgery
Brief Title: Resting-State fMRI Study of Functional Connectivity After Gamma Knife Radiosurgery in Trigeminal Neuralgia
Acronym: DOCTRINE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RCAPHM25_0106_DOCTRINE
Record Dates: First submitted 2026-01-08; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Trigeminal Neuralgia
MeSH Terms: conditions — Trigeminal Neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gamma Knife Radiosurgery - Longitudinal Imaging Follow-up (Experimental)
  Interventions: Procedure: Resting-State Functional MRI

INTERVENTIONS:
Procedure: Resting-State Functional MRI — Participants undergo non-invasive resting-state functional magnetic resonance imaging (rs-fMRI) examinations without contrast injection. Imaging sessions are performed before Gamma Knife radiosurgery and at 1 month, 3 months, and 12 months after treatment. These MRI procedures are conducted solely for research purposes and do not modify standard clinical care. The intervention aims to assess longitudinal changes in brain functional connectivity and their association with clinical outcomes.

SUMMARY:
Trigeminal neuralgia is a severe chronic pain condition with a major impact on quality of life. Although Gamma Knife radiosurgery is an established treatment for pharmacoresistant trigeminal neuralgia, its mechanisms of action and the temporal dynamics of clinical response remain incompletely understood.

This prospective longitudinal study aims to investigate changes in brain functional connectivity using resting-state functional magnetic resonance imaging (rs-fMRI) in patients with classical trigeminal neuralgia treated with Gamma Knife radiosurgery. Participants will undergo rs-fMRI examinations before treatment and at 1 month, 3 months, and 12 months after radiosurgery.

Functional connectivity patterns will be analyzed over time and correlated with clinical outcomes, including pain intensity and treatment response. Imaging data will be compared with those from a cohort of age- and sex-matched healthy volunteers. The study does not modify standard clinical care; only additional non-invasive MRI examinations without contrast injection are performed for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 73 years
* Diagnosis of classical trigeminal neuralgia confirmed by an experienced neurologist
* Unilateral facial pain with a normal neurological examination
* Pharmacoresistant trigeminal neuralgia, defined as failure of at least two appropriate medical treatments, intolerance to medication, or recurrence despite adequate treatment
* Indication for Gamma Knife radiosurgery as part of standard clinical care
* Affiliation to a social security or health insurance system
* Ability to understand the study information and provide written informed consent

Exclusion Criteria:

* Diagnostic uncertainty or secondary/idiopathic trigeminal neuralgia
* Previous surgical or radiosurgical treatment for trigeminal neuralgia
* Participation in another interventional clinical study at the time of inclusion
* Individuals belonging to protected populations as defined by applicable regulations (including minors, adults under legal protection, persons deprived of liberty, pregnant or breastfeeding women)
* Inability to understand the French language
* Contraindication to 3 Tesla MRI, including claustrophobia, presence of pacemaker, defibrillator, metallic prosthesis, or any MRI-incompatible device or foreign body
* Residence distance incompatible with the required follow-up schedule

Ages: 18 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Normalization of resting-state functional connectivity at 3 months | 3 months after radiosurgery
  Percentage of normalization of resting-state functional MRI (rs-fMRI) connectivity patterns at 3 months after Gamma Knife radiosurgery, compared with pre-treatment imaging and with age- and sex-matched healthy control data.

SECONDARY OUTCOMES:
Longitudinal changes in resting-state functional connectivity | Baseline, 1 month, 3 months, and 12 months after radiosurgery
  Percentage of normalization of rs-fMRI connectivity patterns at 1 month, 3 months, and 12 months after Gamma Knife radiosurgery, compared with pre-treatment imaging.
Pain outcome assessed by Barrow Neurological Institute (BNI) Pain Intensity Scale | Baseline, 1 month, 3 months, and 12 months after radiosurgery
  Change in pain status assessed using the Barrow Neurological Institute Pain Intensity Scale

CONTACTS AND LOCATIONS:
Overall Officials: François CREMIEUX, Study Director — Assistance Publique Hopitaux De Marseille

IPD SHARING:
Plan to Share IPD: No